CLINICAL TRIAL: NCT00641303
Title: A Multi-Center Randomized Controlled Double Blind Trial Assessing the Effect of Acupuncture in Reducing Musculoskeletal Symptoms in Breast Cancer Patients Taking Aromatase Inhibitors
Brief Title: Acupuncture in Reducing Muscle and Bone Symptoms in Women Receiving Letrozole, Exemestane, or Anastrozole for Stage 0, Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HP-00043225; P30CA006973 (NIH); JHOC-J07110; SKCCC J07110; JHOC-NA_00013024; GCC 0930 (Other: University of Maryland Greenebaum Cancer Center)
Record Dates: First submitted 2008-03-21; First posted 2008-03-24 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2012-01

CONDITIONS: Anxiety Disorder; Breast Cancer; Depression; Fatigue; Hot Flashes; Pain; Sleep Disorders
Keywords: pain; fatigue; hot flashes; sleep disorders; depression; anxiety disorder; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Depression; Fatigue; Hot Flashes; Pain; Sleep Wake Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (control) (Sham Comparator): Patients receive 8 weekly sessions of sham acupuncture treatment comprising 20 minutes of a non-penetrating device consisting of a retractable needle and an adhesive tube on the skin using the Park Sham Device (PSD) in 14 non-acupuncture points. Patients may receive 4 free acupuncture sessions (not sham) after the 12 or 24-week follow-up visit.
  Interventions: Procedure: sham intervention
- Arm II (treatment) (Experimental): Patients receive 8 weekly sessions of acupuncture treatment comprising 20 minutes of needle insertion in 15 acupuncture points including CV 4, CV 6, CV12 and bilateral LI 4, MH 6, GB 34, ST 36, KI 3, BL 65.
  Interventions: Procedure: acupuncture therapy

INTERVENTIONS:
Procedure: acupuncture therapy — Given weekly for 8 sessions
  Other Names: acupuncture
  Arms: Arm II (treatment)
Procedure: sham intervention — Given weekly for 8 sessions
  Other Names: sham acupuncture
  Arms: Arm I (control)

SUMMARY:
RATIONALE: Acupuncture may help relieve muscle and bone pain caused by aromatase inhibitor therapy, such as letrozole, exemestane, and anastrozole.

PURPOSE: This randomized phase II trial is studying acupuncture to see how well it works in reducing muscle and bone symptoms in women receiving letrozole, exemestane, or anastrozole for stage 0, stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if acupuncture can reduce aromatase inhibitor (AI)-associated musculoskeletal symptom severity, in terms of function and pain, in woman with stage 0-III breast cancer.

Secondary

* To assess if acupuncture decreases oral analgesic use in these patients.
* To assess if acupuncture decreases the proportion of patients who change or discontinue AI therapy.
* To assess if acupuncture improves menopausal symptoms, mood (i.e., depression or anxiety), sleep quality and sleep disturbance, and overall quality of life of these patients.
* To assess if acupuncture changes plasma concentrations of estrogens (i.e., E1, E2, and E1S), cytokine profile, and beta endorphin.

OUTLINE: This is a multicenter study. Patients are stratified according to participation in the aromatase inhibitor trial, "A Multicenter Randomized Clinical Trial Correlating the Effects of 24 Months of Exemestane or Letrozole on Surrogate Markers of Response With Aromatase Polymorphism" (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I (control): Patients receive 8 weekly sessions of sham acupuncture treatment comprising 20 minutes of a non-penetrating device consisting of a retractable needle and an adhesive tube on the skin using the Park Sham Device (PSD) in 14 non-acupuncture points. Patients may receive 4 free acupuncture sessions (not sham) after the 12-week (previously 24-week) follow-up visit.
* Arm II (treatment): Patients receive 8 weekly sessions of acupuncture treatment comprising 20 minutes of needle insertion in 15 acupuncture points including CV 4, CV 6, CV12 and bilateral LI 4, MH 6, GB 34, ST 36, KI 3, BL 65.

Quality of life is assessed periodically to measure changes in symptoms that may be related to hot flashes and estrogen deprivation (i.e., menopausal symptoms, mood [depression and anxiety], sleep quality, and overall quality of life using the menopausal symptoms checklist); the Hot Flash Related Daily Interference Scale (HFRDI) and the Hot Flash Daily Diary; the Pittsburgh Sleep Quality Index (PSQI); the Center for Epidemiologic Studies Depression Scale (CESD); the Hospital Anxiety and Depression Scale (HADS-A); and the EuroQOL.

Patients complete questionnaires including the Health Assessment Questionnaire (HAQ) and visual analog scales (VAS) to assess both pain and global health status at baseline, after 4 and 8 weeks of acupuncture or sham acupuncture, and at follow-up at 12 weeks (previously 24 weeks). The average amount of daily oral analgesic usage is assessed at weeks 0, 4, 8, and 12(previously 24).

Patients undergo blood sample collection periodically for correlative studies. Samples are analyzed for plasma concentrations of estrogen (i.e., estrone E1, estradiol E2, and estrone sulfate E1S) via HPLC-MS/MS, level of 35 serum cytokines via addressable laser bead immunoassay (ALBIA) or classical sandwich ELISA, cytokines and their soluble receptors via classical sandwich ELISA techniques, and Beta-endorphin via competitive ELISA.

All patients are followed for 12 weeks(previously 24 weeks). Patients in arm I may be followed for an additional 4 weeks if they choose to receive the free acupuncture sessions.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive carcinoma of the breast

  * Stage 0-III disease
* Estrogen receptor- and/or progesterone receptor-positive by immunohistochemical staining
* Must be receiving a standard dose of aromatase inhibitor (AI) therapy (i.e., letrozole 2.5 mg once daily, exemestane 25 mg once daily, or anastrozole 1 mg once daily)

  * AI therapy has been ongoing for ≥ 1 month and treatment is expected to continue
* AI-associated musculoskeletal symptoms, defined as ≥ 1 of the following:

  * Physician-confirmed AI-associated musculoskeletal symptoms
  * Patients concurrently enrolled on the clinical trial, "A Multi-Center Randomized Clinical Trial Correlating the Effects of 24 Months of Exemestane or Letrozole on Surrogate Markers of Response with Aromatase Polymorphism," and who have met the referral criteria for a rheumatological evaluation
* No known metastatic (stage IV) breast cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Female
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* No prior acupuncture within past 12 months.
* No other concurrent systemic therapy (i.e., chemotherapy, biologic therapy, or radiotherapy) unless approval is given by the Protocol Chair

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-05; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Health Assessment Questionnaire Disability Index (HAQ-DI) score | Baseline, Weeks 4, 8 and 12 (or Week 24)
Pain scores on visual analog scale (VAS) | Baseline, Weeks 4, 8 and 12 (or Week 24)

SECONDARY OUTCOMES:
Change in amount and/or frequency of oral analgesic use | Baseline, Weeks 1-8, Week 12 (or Week 24)
Number of patients who discontinue or change AI therapy | All timepoints
Change in menopausal symptoms (NSABP-revised), hot flash frequency (HFRDIS), sleep quality (PSQI), depression score (CESD), and overall quality of life (EuroQOL) in patients at weeks 4, 8, and 24 vs week 0 of acupuncture treatment | Baseline, Weeks 4, 8 and 12 (or Week 24)
Change in plasma estrogen concentrations, beta endorphin concentration, and cytokine profile from week 0 to week 8 | Baseline, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, Principal Investigator — University of Maryland Marlene & Stewart Greenebaum Cancer Center
Locations (2):
- United States (2):
  - University of Maryland Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland